

黄偉國教授 Professor Rick W. K. Wong PhD, MSc (DIC) Chair Professor in Chemistry

29 April 2016

Dr. Duan Yanping

PE

Dear Dr. Duan,

# Re: The Effectiveness of an E-Intervention on Health Behavior Promotion for Chinese University Students [FRG2/15-16/032]

I refer to your application for a Faculty Research Grant.

The Arts and Social Sciences Specialist Panel, a subcommittee of the Research Committee, has recently considered the above proposal and resolved that a research grant in the amount of **HK\$150,000.00** be awarded in support of the proposal. Details of the grant are specified on the attached sheet (*Form RC/01a*). Please quote the number code of the project in all future correspondence and requisition/reimbursement requests.

The expected completion date for the above project is **31 December 2017**. Please submit an online completion report via the Research Project System through the BUniPort to the Research Committee **within 6 months from that date**. Should you encounter any difficulties in meeting the deadline, a progress report together with a request for extending the deadline should be forwarded to the Chairman of the Research Committee for consideration prior to the due date. In addition to the completion report, the Committee also reserves the right to request a progress report from you at times deemed appropriate.

On behalf of the Research Committee, I wish you every success in bringing your project to a fruitful conclusion.

Yours sincerely,

Prof. Rick W. K. Wong

Chairman

Research Committee

cc Dean, SOSC Head/Director, PE Finance Office Personnel Office Library (RVP Team)

Encl.

**Note:** Please refer to para. 10 of the attached Form RC/01a "Conditions/Information on Research Grant Approval" for downloading of relevant guidelines and forms pertaining to the grant

## **Faculty Research Grant**

## Conditions/Information on Research Grant Approval

1. Project no.: FRG2/15-16/032

2. Title of project: The Effectiveness of an E-Intervention on Health Behavior Promotion

for Chinese University Students

3. Principal Investigator: Dr. Duan Yanping, PE

4. Co-investigator(s): Mr. Chen Xu, Department of Physical Education,

Nantong University, P.R. China

Dr. Cui Degang, Physical Education Section, Wuhan

University, P.R. China

Dr. Lin Zhihua, Physical Education Section, Wuhan

University, P.R. China

Prof. Lippke Sonia, Jacobs Center on Lifelong Learning

and Institutional Development, Jacobs University

Bremen, Germany

5. Duration of project: From 1 June 2016 to 31 December 2017

6. Funding approved:

Total allocation: HK\$150,000

7. Breakdown of proposed budget items:

| Item | Estimated Expenditure |
|------|-----------------------|
| | (HK\$) |

Staff

7.1 Research Assistant \$109,080

\$10,908 x 10 months

**General Expenses** 

7.2 Website set-up (\$18,000) \$30,920

Promotional materials (\$3,000)

Transportation and accommodation expenses (\$9,920)

Conference Cost

7.3 Conference and publication charges \$10,000

Total \$150,000

#### 8. Procedures to observe:

- 8.1 The reading materials purchased through the allocated funding will need to be returned to the Faculty/School/Academy on completion of the project and subsequently catalogued and retained by the University library.
- 8.2 Reimbursement/purchase requisition forms: Unless otherwise authorized, these forms should be signed by the Principal Investigator (PI) who is the only person in the team authorized to sign such requests. In the event of the PI being absent from the University for a lengthy period, the team may wish to consider appointing a temporary deputy to submit requests. The Graduate School and the Finance Office should be notified of such arrangements prior to the commencement of the leave period of the PI. Requests signed by team members other than the PI will normally be considered null and void by the Finance Office.

## 9. Remarks/Conditions:

- 9.1 Corruption Department Independent The Prevention of the Commission Against Corruption (ICAC) advises that Principal Investigators should be reminded of the need to adopt the principles of openness and fairness in matters relating to the research projects especially the recruitment of research staff. In making these appointments, as in the making of all other University appointments which would involve a formal recruitment process to ensure objectivity and impartiality, Investigator are reminded of any likely conflict of interest arising from employing friends or relatives in the same office to avoid any possible suspicion of favouritism or nepotism.
- 9.2 Starting from January 2009, requests for changes such as extension request and submission of completion report should be done by the PI via the Research Project System through the BUniPort.
- 9.3 The proposal may be subject to the approval of the Committee on the Use of Human and Animal Subjects in Teaching and Research (HASC). The Research Committee reserves the right to discontinue funding of this project should the Principal Investigator and Co-investigator(s) (if any) fail to comply with the recommendations/suggestions of HASC.
- 9.4 As approved by the Research Committee on its 2nd meeting 2014/15, academic colleagues, who have been awarded internal grants or matching support from the Research Committee, are required to participate the Research Visibility Project (RVP) which is administered by the Library.

NOTE:

10. Relevant guidelines and forms can be downloaded from the Graduate School website below:

http://gs.hkbu.edu.hk/en/staff/grants/login staff&restricted

#### INFORMED CONSENT STATEMENT (for Fast Track Review)

#### STUDY INFORMATION SHEET

[The Effectiveness of an E-Intervention on Health Behavior Promotion for Chinese University Students]

- ---You are invited to participate in a research study. The purpose of this study is to provide you an innovative e-health learning program targeting physical activity and dietary behaviour, which you can follow in your spare time. The outcomes of this research project will provide knowledge relative to:
- 1. Examining whether the participants are able to gain a higher motivation for physical activity and healthy dietary by participating in this program.
- 2. Examining whether participants in the intervention groups increase their physical activity levels and healthy diet consumption compared to the control group.
- 3. Examining whether the intervention program can improve participants' perceived quality of life.

## **INFORMATION**

Participating in this study, you will receive an eight-week intervention after you discharge from rehabilitation. You are required to access to an e-health website once per week during this program period. Each e-learning session will cost approximately 15 minutes in average. The internet website contains several learning modules, such as information pages regarding how to engage in appropriate physical activity and maintain healthy dietary, digital personalized agenda in which you formulate your activity plans, nutrition plans, as well as health model learning to increase your motivation and self-confidence on physical activity and nutrition. Besides, you will be further contacted for collecting data at the beginning of intervention (T1), at the end of intervention (T2), and 1 month after the intervention (T3).

Each electronic questionnaire survey will last approximately 15 minutes. All information you provided will be kept strictly confidential. Only the results of statistical analyses will be reported. Please indicate your true perception or feeling about issues described in the questionnaire.

#### BENEFITS

You will obtain supporting information about physical activity and dietary behaviour by the way of e-health learning in your spare time, in the long-term, which might not only maintain the intention, increase planning, coping abilities and well-being, but might also keep you fit by means of implementing healthy behavior habit.

## **CONFIDENTIALITY**

As this study will be conducted over the internet, we cannot guarantee confidentiality while your data is on the internet. In addition, the identifiers will be destroyed within 6 months upon the completion of this study.

#### COMPENSATION AND INSURANCE

For participants in this project, you will be offered RMB 45 mobile charge as incentive immediately after the completion of this study. If you withdraw from the study prior to its completion, you won't receive it.

#### **CONTACT**

If you have questions at any time about the study or the procedures, you may contact the researcher, Dr. Duan Yanping at 852-34113080 or <a href="duanyp@hkbu.edu.hk">duanyp@hkbu.edu.hk</a>. If you feel you have not been treated according to the descriptions in this form, or your rights as a participant in research have been violated during the course of this project, you may contact the Committee on the Use of Human and Animal Subjects in Teaching and Research by email at <a href="hasc@hkbu.edu.hk">hasc@hkbu.edu.hk</a> or by mail to Graduate School, Hong Kong Baptist University, Kowloon Tong, Hong Kong.

## **PARTICIPATION**

(Applied for students under 18)

Your participation in this study is voluntary; you may decline to participate without penalty. If you decide to participate, you may withdraw from the study at any time without penalty and without loss of benefits to which you are otherwise entitled. If you withdraw from the study before data collection is completed your data will be returned to you or destroyed.

## **CONSENT**

| Signature of the Subject | Date |
|-------------------------------------------------------|------|
| Signature of Parents(s)/Guardian/Legal Representative | Date |

I have read and understand the above information. I have received a copy of this form. I agree to participate in this study.

| Signature of the Investigator | Date |
|-------------------------------|------|

# 同意書 - 適用於簡易審核

## 【中国大学生网络学习健康促进效益研究】

---您受邀参加这项研究。该研究旨在<u>以网络学习的方式促进体育运动和饮食健康行为,整个过程是</u> 在您学业之余完成的。研究目的包括以下四个方面:

- 1. 探究项目参与者在体育运动和饮食健康两方面的动机是否有所提高。
- 2. 探究网络健康学习是否有助于增加参与者的运动量和健康饮食摄入量。
- 3. 探究网络健康学习是否有助于提升参与者的生活质量感。

## 背景资料

整个研究是在您的业余时间完成的。我们为您提供为期8周的(网络健康学习)干预方案,在整个过程中,您需要每周一次上网浏览我们制作的网络健康学习网站,每次大约耗用您15分钟。该网站包括许多学习模块,在"信息"页面您可以获悉如何参加体育运动,如何保持饮食健康;在"网络个人日程"里您可以为体育运动和饮食健康制定计划,在"健康"页面,您可以学习到如何提高(体育运动和饮食健康方面的)动机和自信水平。除了上述内容,您需要在我们的网络健康网站上完成3次网络问卷,施测时间分别为干预之初(T1),干预结束后(T2),以及干预结束一个月之后(T3)。

每份网络问卷耗时大约 15 分钟,我们会对您填写的所有信息进行保密,只会发表统计分析的结果,所以请您真实的完成问卷。

## 研究效益

您可以在业余时间以网络学习的方式获得有关于体育运动和饮食健康行为的信息,从长远角度而言,这不仅可以帮助您保持(体育运动和健康饮食的)行为意愿;提高您制定计划、实施计划的能力;还可以帮助您通过实施健康的行为习惯保持健康状态。

## 隐私保障

由于本研究将通过网络进行,对于您在网络上填写的信息,我们将无法完全保证数据的保密性。此外,所有收集到的信息将会在研究结束后的六个月内全部销毁。

# 补偿方式

如果您参与本项目,您将在研究结束后立即获得 45 元的手机充值话费作为奖励。如果您中途退出, 将无法获得此待遇。

# 联络资料

如果您对本研究有任何疑问,请联系段艳平博士,电话: +852 3411 3080,邮箱: duanyn@hkbu edu hk 如果您在参与研究的过程中发现实际情况与本文件所述内容不

duanyp@hkbu.edu.hk。如果您在参与研究的过程中发现实际情况与本文件所述内容不相符,或者感到自己作为参与者的权益受到侵犯,请您以网络邮件的方式(hasc@hkbu.edu.hk)与教研所用人畜实验监管委员会联系,或者写信给香港浸会大学研究生院。

# 参与条款

| 您是否参与本研究是完 | 全自愿的, | 拒绝参与不 | 一会受到任何惩罚 | 引。中途 | 退出不会 | 受到惩罚, | 所享有的 |
|------------|-------|-------|----------|------|-------|-------|------|
| 权益也不会受到损害。 | 如果您在對 | 据收集结束 | 之前决定退出本 | 体研究, | 那您的数据 | 居将会被退 | 还或者销 |
| 毁。 | | | | | | | |

| $\rightarrow$ | | - 1 |
|---------------|---------------|-----|
| | <del>~~</del> | - |
| ΙПΙ | | |
| I, A | VEV. | 14 |

我已经阅读了上述研究信息。我同意参加该项研究。

| 参与者: | 日期 |
|---------------------------------|----------|
| 监护人:<br>(活用工 10 出以工 <u>类</u> 集) | 日期 |
| (适用于 18 岁以下学生) | No. |
| 调查者: | _ 日期 |